CLINICAL TRIAL: NCT06585371
Title: Evaluation of the Safety and Efficacy of a 6-month Intragastric Balloon
Brief Title: Evaluation of a 6-month Intragastric Balloon
Status: Not yet recruiting | Type: Observational
Sponsor: MEDICONE PROJETOS E SOLUCOES PARA A INDUSTRIA E A SAUDE LTDA (Other)
Responsible Party: Sponsor
Other Study IDs: MEDICONE_01_2024
Record Dates: First submitted 2024-08-28; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Obesity and Overweight
Keywords: intragastric; weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with intragastric balloon: Patients over 18 years old, who are overweight, have a BMI of 27 kg/m2 or greater and are going through intragastric balloon placement.

SUMMARY:
Post-market observational, adaptive, single-arm clinical study to evaluate the percentage of total weight loss after treatment with an intragastric balloon. Patients will be followed for 6 months after the device is installed.

DETAILED DESCRIPTION:
Forty-six overweight patients over 18 years of age with a BMI of 27 kg/m2 or greater who are considered suitable for intragastric balloon placement will be included. The primary outcome will be the assessment of the percentage of total weight loss (%WL) at 6 months. Patients will be screened in an outpatient setting at the participating research center. All participants who meet the eligibility criteria will be invited to participate in the study, which includes a screening visit, standard intragastric balloon placement procedure, and follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Age 18 or older;
* Both sexes;
* Being overweight, with a Body Mass Index (BMI) of 27 kg/m2 or higher;
* Being able to follow the protocol monitoring requirements;
* Adhering to the diet recommended by the nutrition professional;
* Presenting reasonable expectations of weight loss, at least 10% of baseline weight.

Exclusion Criteria:

* Pregnant women or women during the breastfeeding period;
* People unable or unwilling to comply with restrictions regarding diet or medical monitoring and their respective guidelines during the program for use of the Intragastric Balloon;
* People with severe kidney and/or liver diseases;
* Patients who have undergone previous gastric surgery;
* Patients with inflammatory diseases of the gastrointestinal tract, gastric ulcer, duodenal ulcer or specific inflammations, such as Crohn's disease, or with a propensity for gastrointestinal bleeding in the upper tract, such as esophageal or gastric varices, or acquired intestinal telangiectasia;
* People with severe cardiopulmonary or organic disorders;
* People with congenital or acquired anomalies of the gastrointestinal tract, such as atresia and stenosis; with large hiatal hernia;
* Drug addicts in general;
* Patients not committed to adhering to treatment and medical recommendations, including nutritional guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who are overweight, with a Body Mass Index (BMI) of 27 kg/m2 or greater and who are considered fit to undergo the procedure for placement of the intragastric balloon
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the percentage of total weight loss (%PPT) in 6 months after installation of the intragastric balloon | From the installation of the balloon to the end of treatment at 6 months
  To analyze the percentage of total weight loss 6 months after installation of the intragastric balloon, the following formula will be used:
  Percentage of total weight loss = kilos lost/initial weight x 100

SECONDARY OUTCOMES:
Number of Adverse event occurrence assessed by clinical evaluation | From the installation of the balloon to the end of treatment at 6 months
  Adverse event monitoring through medical clinical evaluation
Weight changes 6 months after installation of the balloon assessed by anthropometric balance in in-person consultations | From the installation of the balloon to the end of treatment at 6 months
  Patients will be weighed on an anthropometric balance during in-person consultations
BMI changes 6 months after the installation of the intragastric balloon assessed by BMI calculation in in-person clinical consultations | From the installation of the balloon to the end of treatment at 6 months
  To analyze the BMI changes, the BMI will be calculated in the follow-up medical consultations by dividing the weight (in kg) by the square of the height (in meters), according to the following formula: BMI = weight/(height x height)
Abdominal circumference changes 6 months after the intragastric balloon installation assessed by measuring tape in in-person clinical consultations | From the installation of the balloon to the end of treatment at 6 months
  To measure abdominal circumference, during in-person medical consultations, the patient will stand with arms extended at the side of the body, feet apart and parallel. The measuring tape will be positioned around the abdomen, midway between the lower costal margin and the iliac crest.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kolotkin RL, Meter K, Williams GR. Quality of life and obesity. Obes Rev. 2001 Nov;2(4):219-29. doi: 10.1046/j.1467-789x.2001.00040.x. PMID 12119993
- [Background] Caballero B. Humans against Obesity: Who Will Win? Adv Nutr. 2019 Jan 1;10(suppl_1):S4-S9. doi: 10.1093/advances/nmy055. PMID 30721956
- [Background] Lee KG, Nam SJ, Choi HS, Lee HL, Yoon JH, Park CH, Kim KO, Kim DH, Kim JW, Sohn W, Jung SH; Korean Research Group for Endoscopic Management of Metabolic Disorder and Obesity. Efficacy and safety of intragastric balloon for obesity in Korea. Clin Endosc. 2023 May;56(3):333-339. doi: 10.5946/ce.2022.143. Epub 2022 Dec 13. PMID 36510655
- [Background] Martinez-Brocca MA, Belda O, Parejo J, Jimenez L, del Valle A, Pereira JL, Garcia-Pesquera F, Astorga R, Leal-Cerro A, Garcia-Luna PP. Intragastric balloon-induced satiety is not mediated by modification in fasting or postprandial plasma ghrelin levels in morbid obesity. Obes Surg. 2007 May;17(5):649-57. doi: 10.1007/s11695-007-9109-z. PMID 17658025
- [Background] Genco A, Cipriano M, Bacci V, Cuzzolaro M, Materia A, Raparelli L, Docimo C, Lorenzo M, Basso N. BioEnterics Intragastric Balloon (BIB): a short-term, double-blind, randomised, controlled, crossover study on weight reduction in morbidly obese patients. Int J Obes (Lond). 2006 Jan;30(1):129-33. doi: 10.1038/sj.ijo.0803094. PMID 16189503
- [Background] Guedes EP, Madeira E, Mafort TT, Madeira M, Moreira RO, Mendonca LM, Godoy-Matos AF, Lopes AJ, Farias ML. Impact of a 6-month treatment with intragastric balloon on body composition and psychopathological profile in obese individuals with metabolic syndrome. Diabetol Metab Syndr. 2016 Dec 19;8:81. doi: 10.1186/s13098-016-0197-6. eCollection 2016. PMID 28031749
- [Background] Buzga M, Evzen M, Pavel K, Tomas K, Vladislava Z, Pavel Z, Svagera Z. Effects of the intragastric balloon MedSil on weight loss, fat tissue, lipid metabolism, and hormones involved in energy balance. Obes Surg. 2014 Jun;24(6):909-15. doi: 10.1007/s11695-014-1191-4. PMID 24488758
- [Background] Moore RL, Eaton L, Ellner J. Safety and Effectiveness of an Intragastric Balloon as an Adjunct to Weight Reduction in a Post-Marketing Clinical Setting. Obes Surg. 2020 Nov;30(11):4267-4274. doi: 10.1007/s11695-020-04798-5. PMID 32617919